CLINICAL TRIAL: NCT06208969
Title: Comparison of Intensive and Standard Nutrition Counseling in Monitoring the Nutritional Status of Stroke Patients
Brief Title: The Effect of Nutrition Counseling on Nutritional Status in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Dilek Seyidoglu Yuksel, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-3.1T/14
Record Dates: First submitted 2023-12-02; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute; Malnutrition; Old Age; Debility
Keywords: malnutrition; older
MeSH Terms: conditions — Stroke; Malnutrition; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensive nutrition counseling (Experimental): Five-stage nutrition counseling vith educational materials was carried out during hospitalization in the intensive nutrition counseling. Telephone interviews were conducted at the 2nd week and 2nd month after discharge.
  Interventions: Behavioral: intensive nutrition counseling
- standard nutrition counseling (Active Comparator): Routine nutritional counseling was applied. Interviewed only at admission and at discharge if patient is consulted.
  Interventions: Behavioral: intensive nutrition counseling

INTERVENTIONS:
Behavioral: intensive nutrition counseling — individualized regular nutrition education

SUMMARY:
The purpose of this study is to investigate the effect of intensive nutrition counseling on nutritional status and functional recovery in stroke patients over the age of 65, compared to standard nutrition counseling.

DETAILED DESCRIPTION:
Stroke is the second most common cause of death in the world; It is the third cause of disability that causes serious loss of function and affects patients' daily activities. The rapid aging of society increases the negative impact of stroke on health and limited health resources. 9-35% of patients hospitalized with the diagnosis of acute stroke have malnutrition. However, in the first two weeks after hospitalization, malnutrition rates approximately double within two weeks of hospitalization. Although nutrition is a physiological need, it is also a social activity. Nutritional practices that meet nutritional needs during the disease process may contribute to the functional recovery of patients, the reduction of complications, and survival, as well as contributing to the quality of life of patients, independent of the disease. In terms of malnutrition risk, monitoring and treatment are recommended during the acute and discharge periods. There is a need for studies on the framework and effects of effective nutritional treatment. In order for nutrition treatment practices after discharge to achieve their goals, caregivers need to be trained effectively on this subject. Therefore, the aim of this study is to examine the effects of intensive nutrition counseling to stroke patients over the age of 65 on nutritional and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Being admitted to Ege University Faculty of Medicine Hospital Neurology Intensive Care or Clinic with the diagnosis of acute stroke
* The patient agrees to participate in the study
* Hospital stay for more than 3 days

Exclusion Criteria:

* Active malignancy, dementia, terminal illness, tetraplegia, severe metabolic disorder
* Failure to obtain written consent indicating that they agreed to participate in the study.
* The patient did not come for a check-up during the 3-month follow-up period
* The patient's stay is longer than 30 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — over 65 years old
Enrollment: 61 (Actual)
Dates: Start 2021-03-07 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Malnutrition Risk | Hospitalization (up to day 5), first month after discharge, third month after discharge
  Malnutrition risk status according to MUST
BMI | Hospitalization (up to day 5), first month after discharge, third month after discharge
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. If BMI<22 kg/m2, it is considered low
Calf Circumference Measurement | Hospitalization (up to day 5), first month after discharge, third month after discharge
  The widest part of the calf was measured from the non-paralyzed side in a sitting position with 90 degrees.
Malnutrition | Hospitalization (up to day 5), first month after discharge, third month after discharge
  Malnutrition diagnosis according to GLIM criteria
Mid Upper Arm Circumference | Hospitalization (up to day 5), first month after discharge, third month after discharge
  Mid upper arm circumference is measured at the midpoint between the acromion and olecranon processes on the shoulder blade and the ulna.
Mid Upper Arm Muscle Area | Hospitalization (up to day 5), first month after discharge, third month after discharge
  Mid upper arm muscle area is calculated using the standard formula= Mid Upper Arm Circumference-(3.14 x Triceps skinfold thickness)

SECONDARY OUTCOMES:
Functional Status | last day of hospitalization, first month after discharge, third month after discharge
  Functional status was evaluated according to the Barthel Activities of Daily Living İndex
Disability | last day of hospitalization, first month after discharge, third month after discharge
  Disability was evaluated according to The Modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sevnaz Sahin, Assoc Prof, Study Director — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided